CLINICAL TRIAL: NCT01056419
Title: The Effect of Early Total Thyroidectomy in the Course of Graves' Orbitopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ankara University (Other)
Responsible Party: Ankara University, Medical School, Ankara University, Medical School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08067
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2009-06

CONDITIONS: Graves' Ophthalmopathy
Keywords: Graves' ophthalmopathy; Total thyroidectomy; Anti-thyroid drug treatment; Clinical activity score
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Propylthiouracil

ARMS (2):
- Total thyroidectomy (Active Comparator)
  Interventions: Procedure: Total Thyroidectomy
- Anti-thyroid drug (Active Comparator)
  Interventions: Drug: Propylthiouracil

INTERVENTIONS:
Procedure: Total Thyroidectomy — Total thyroidectomy within 6 months after the appearance of the symptoms of ophthalmopathy
  Arms: Total thyroidectomy
Drug: Propylthiouracil — 150-600 mg in two-three divided doses
  Arms: Anti-thyroid drug

SUMMARY:
The relationship between the method of the treatment of hyperthyroidism due to Graves' disease and the course of Graves' ophthalmopathy is debated. The investigators aimed to compare the results of total thyroidectomy done in 6 months following the appearance of the symptoms of ophthalmopathy and the antithyroid drug therapy in patients with moderate to severe Graves' ophthalmopathy.

The inclusion criteria: 1)Hyperthyroidism and moderate to severe Graves' ophthalmopathy within 6 months, 2)Thyroid volumes greater than or equal to 15 mL in thyroid ultrasonography, 3)Patients taking no treatment except local medications for Graves' ophthalmopathy, 4)Clinical activity score of 3/7 or more, proptosis greater than or equal to 21 mm in one eye or 2 mm difference between two eyes, presence of diplopia, the opening of the eye lid greater than or equal to 9 mm.

All patients will be treated with antithyroid drug until TSH levels of the patients are between 0.4-1. During this period all the patients will take pulse methyl prednisolone treatment of a total dose of 4.5 gr. After pulse steroid treatment the patients will be randomised to two groups: one group will be sent to surgery for total thyroidectomy, and their TSH levels will be kept between 0.4-1 with levothyroxine treatment; the other group will be followed under antithyroid drug treatment and their TSH levels will be kept between 0.4-1 also.

The smoking habits will be asked. Serum TSH, fT4 levels, Hertelmeter and eye lid opening measurements, clinical activity scores, diplopia will be evaluated monthly; TSH receptor antibody, anti-thyroid peroxidase and anti-thyroglobulin levels will be measured in 3 months intervals for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Hyperthyroidism and moderate to severe Graves' ophthalmopathy within 6 months,
* Thyroid volumes greater than or equal to 15 mL in thyroid ultrasonography,
* Patients taking no treatment except local medications for Graves' ophthalmopathy,
* Clinical activity score of 3/7 or more, proptosis greater than or equal to 21 mm in one eye or 2 mm difference between two eyes, presence of diplopia, the opening of the eye lid greater than or equal to 9 mm.

Exclusion Criteria:

* Patients taking treatment other than local medications for Graves' ophthalmopathy (eg: steroid treatment)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-06 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Improvement in the proptosis and activity of Graves' ophthalmopathy | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Medical School, Ibni Sina Hospital, Endocrinology and Metabolic Diseases Department, Ankara, Turkey (Türkiye)